CLINICAL TRIAL: NCT03311295
Title: MitrAl ValvE RepaIr Clinical Trial (MAVERIC Trial) - United States
Acronym: MAVERIC US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lagging enrollment
Sponsor: Mvrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US042616
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ARTO System (Experimental)
  Interventions: Device: ARTO System

INTERVENTIONS:
Device: ARTO System — The ARTO System directly reshapes the mitral annulus promoting leaflet coaptation and amelioration of regurgitation.

SUMMARY:
The objective of the study is to evaluate the safety and feasibility of the ARTO System in patients with mitral valve regurgitation (MR) associated with congestive heart failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

Candidates must meet ALL of the following criteria to be enrolled in the study.

* Is ambulatory, able and willing to comply with the study protocol and has provided written informed consent
* Age 21-85, inclusive
* Trans-septal catheterization is determined to be feasible by the treating physician
* NYHA class II-IV heart failure of any etiology
* Symptomatic with MR grade ≥ 2+
* LVEF < 40%
* LVEDD > 50 mm and ≤ 75 mm
* No anticipated change in patient's cardiac medication regimen anticipated throughout the course of the study.
* In the opinion of the investigator and heart surgery team, the patient is not an appropriate candidate for surgery, and the use of the ARTO System is technically feasible

Exclusion Criteria:

Candidates will be excluded from enrollment in the study if ANY of the following conditions apply.

* In the opinion of the Investigator, the femoral vein and internal jugular vein cannot accommodate a 16 F catheter or the presence of an inferior vena cava (IVC) filter would interfere with advancement of the catheter or ipsilateral DVT is present
* Significant structural abnormality of the mitral valve (e.g., flail, prolapse, leaflet calcification)
* Significant mitral annular calcification
* Hemodynamic instability (systolic pressure < 90 mmHg without afterload reduction or cardiogenic shock or the need for inotropic support or intra-aortic balloon pump)
* Prior mitral valve surgery or valvuloplasty or any currently implanted prosthetic valve or VAD
* History of, or active, rheumatic heart disease
* History of Atrial Septal Defects (ASD), whether repaired or not
* History of previously repaired PFO or PFO associated with clinical symptoms (e.g., cerebral ischemia) within 6 months of the planned investigational procedure
* In the opinion of the investigator, an atrial septal aneurysm is present that may interfere with transseptal crossing
* Serum creatinine > 2.5 mg/dL or dialysis dependent
* No access to coronary sinus and/or great cardiac vein
* Platelet count < 100 x 103 cells/mm3
* Evidence of active infection (fever with temperature > 38°C and/or WBC > 15,000) or endocarditis
* Echocardiographic evidence of mass intracardiac thrombus
* Patients on prescribed dual antiplatelet therapy (asprin + any P2Y12 inhibitor) that cannot be discontinued.
* Percutaneous coronary intervention or surgery anticipated within the 6 month follow up period following the investigational procedure
* Biventricular pacing initiated or anticipated within 6 months of the planned investigational procedure
* Evidence of an acute myocardial infarction within 12 weeks of the planned investigational procedure
* Stroke or TIA within 6 months of the planned investigational procedure
* GI bleeding within 6 months of the planned investigational procedure
* Intravenous drug abuse or suspected inability to adhere to follow-up
* Patients in whom TTE, TEE or ICE is contraindicated
* Contraindication to CT scan
* A known hypersensitivity or contraindication to study or procedure medications (specifically aspirin, clopidogrel and heparin) that cannot be adequately managed medically
* A known allergy or hypersensitivity to nickel
* A known need for any other cardiac surgery including surgery for coronary artery disease, atrial fibrillation, pulmonic, aortic or tricuspid valve disease
* In the judgment of the Investigator, patients in whom the presence of a permanent pacemaker or pacing leads would interfere with placement of the test device or the placement of the test device would disrupt the leads
* Irreversible bleeding disorder, history of bleeding diathesis or coagulopathy or refuses blood transfusion
* Evidence of disease or condition expected to compromise survival (< 1 year) or ability to complete follow-up assessments
* Pregnant or breastfeeding women
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. [Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials]
* Patient not a candidate for emergent surgical bailout in case of need

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Safety: Major Adverse Event Rate to 30 Days post-procedure | 30 days post procedure
  Major Adverse Events (MAEs) will be categorized and defined in accordance with the relation to the procedure and device.
Efficacy: Mitral regurgitation grade by ASE criteria and change from baseline to 1 year | Baseline to 1 year
  Mitral regurgitation grade by ASE criteria and change from baseline to 1 year evaluated by 2-D transthoracic echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Low, MD, Principal Investigator — University California Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States